CLINICAL TRIAL: NCT04847934
Title: Effect Of Distraction Methods On Procedure-Related Fear, Anxiety, And Pain During Intramuscular Injection in Pediatric Emergency Department
Brief Title: Effect Of Distraction Methods On Procedure-Related Fear, Anxiety, And Pain During Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Dokuz Eylul University, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5856-GOA
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-07

CONDITIONS: Pain; Fear; Anxiety; Child, Only
Keywords: intramuscular injection; distraction methods; cold vibration; manuel pressure vibration; virtual reality
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality Group (Experimental): watching the application by wearing virtual glasses to the child during the intramuscular injection
  Interventions: Behavioral: distraction methods
- Manual Pressure Vibration Technique Group (Experimental): Application of manual pressure vibration technique to the area where the intervention will be made
  Interventions: Behavioral: distraction methods
- Cold Vibration Group (Experimental): Buzzy, connecting and operating 5 cm above the area to be injected
  Interventions: Behavioral: distraction methods
- Control Group (No Intervention): Standart care

INTERVENTIONS:
Behavioral: distraction methods — distraction methods
  Arms: Cold Vibration Group; Manual Pressure Vibration Technique Group; Virtual Reality Group

SUMMARY:
Buzzy, shot-blocker, distraction cards, and balloon blowing can reduce fear and pain during the intramuscular intervention in the pediatric emergency service unit. This study aimed to evaluate the effect of virtual reality, manual pressure vibration technique, and cold vibration device application on procedure-related pain, fear, and anxiety during intramuscular antibiotics in children aged 5-12 years in the pediatric emergency department.

DETAILED DESCRIPTION:
Study Hypothesis The pain, fear, and anxiety scores of the children who watch videos with virtual reality glasses during the intramuscular intervention are lower than the other groups.

The pain, fear, and anxiety scores of children who were applied manual pressure vibration technique during the intramuscular intervention are lower than the other groups.

The pain, fear, and anxiety scores of the children who were applied cold vibration (Buzzy) during the intramuscular intervention were lower than the other groups.

The emotional appearance scores of the children in groups before the procedure affect the pain, fear, and anxiety they experience.

The group with children affects the vital signs before and after the distraction technique.

Methods Study Design and Sample It was planned to include children between the ages of 5-12 who will be administered intramuscular antibiotics in the Dokuz Eylül University Pediatric Emergency Service. It is planned to include patients selected by the stratified randomization method in accordance with the sampling criteria.

Randomization Children will allocate by the stratified randomization; gender, age, and antibiotics type. Randomization was performed with a computerized random-number generator.

Socio-Demographic Data Collection and Procedure Follow-up Form: It includes "age, gender, the reason for admitting to the emergency unit, the last painful intervention and date, the name of the antibiotic administered, and the accompanying parent". At the same time, the duration and vital signs of the interventions applied to the child will be recorded.

Wong-Baker FACES (WBS) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity, ranges from 0 (very happy/no pain) to 10 (hurts worst).

The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater response indicates the level of fear. It can be used during the procedure for children aged 5-10 years.

The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety.

Emotional Appearance Scale for Children: This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'.

Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors.

Data collection process Each patient included in the study will be taken to the bed where the intervention will be made and monitored, pulse, respiration, and blood pressure will be measured. The child will be evaluated by the nurse before the procedure with the Emotional Appearance Scale for Children (0. Min).

In the virtual glasses group, the video will be started by wearing virtual glasses.

The manual pressure vibration technique will be applied for 15 seconds. In the cold vibration group, Arı Buzzy will be connected 5 cm above the IM intervention area and applied for 15 seconds.

The hour/minute applied by the IM intervention will be recorded. When he enters the vascular access, he will give information to the child by saying "now it will be over, I am pressing it with cotton". The patient's pulse, respiration, blood pressure will be measured again (minutes will be recorded). Pulse, respiration, and blood pressure will be re-evaluated at the 5th minute of the beginning of the procedure. At the 5th minute of the procedure, the child will be asked to evaluate the most painful moment he feels during the procedure with the Facial Expressions Rating Scale. The child will be given the Child Fear Scale (CAS) and the Child Anxiety Scale-Statefulness (CAS-D) to evaluate how anxious and afraid he or she is during the procedure. You will be asked to mark it with a pencil.

Ethics Ethical approval was received from the Non-Invasive Clinical Studies Ethics Committee of the University where the research was conducted (5856GOA 2021). The researcher informed about the aim of the study and obtained written consent forms from children and parents.

ELIGIBILITY:
Inclusion Criteria:

* Children are between the ages of 5-12
* Intramuscular antibiotics (penicillin, ceftriaxone, amikacin etc.) to be administered
* The intervention will be applied from the gluteal region
* The child agrees to voluntarily participate in the study.
* Parents agree to voluntarily participate in the study
* Obtaining consent form from the child and parent

Exclusion Criteria:

* child with a physical and psychological deficit to prevent him from wearing the glasses to be worn on his head so that he can watch virtual reality.
* child with sedative or analgesic medication.
* child with a neurodegenerative disease, mental retardation, vision and hearing problems, chronic, life-threatening (sepsis, shock, respiratory / cardiac arrest) or genetic disease

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | procedure (during the ıntramuscular injection)
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Anxiety assesed by Children Anxiety Meter-State | procedure (during the intramuscular injection)
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Fear assesed by Child Fear Scale | procedure (during the ıntramuscular injection)
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear. It can be used during the procedure for children aged 5-10 years.

SECONDARY OUTCOMES:
Emotional Appearance Scale for Children | Baseline (before the intramuscular injection)
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'.
  Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Ö Gerçeker, Study Director — RN, PhD, Assoc. Prof.
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulduran E, Ozalp Gerceker G. Effect of Distracting Methods on Procedure-Related Fear, Anxiety, and Pain During Intramuscular Injection: A Randomized Controlled Trial. J Emerg Nurs. 2026 Jan;52(1):127-142. doi: 10.1016/j.jen.2025.08.003. Epub 2025 Sep 9. PMID 40923961